CLINICAL TRIAL: NCT02542943
Title: A Clinical Study Investigating the Efficacy of Two Experimental Oral Rinses in Providing Long Term Relief From Dentinal Hypersensitivity
Brief Title: Efficacy of Two Experimental Oral Rinses in Providing Long Term Relief From Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204762
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental Oral Rinse1 (Experimental): Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 ml of Experimental Oral Rinse 1 for 1 minute. This regimen will be performed twice daily for 8 weeks.
  Interventions: Device: Experimental Oral Rinse 1; Drug: Standard fluoride toothpaste
- Experimental Oral Rinse 2 (Experimental): Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 ml of Experimental Oral Rinse 2 for 1 minute. This regimen will be performed twice daily for 8 weeks.
  Interventions: Device: Experimental Oral Rinse 2; Drug: Standard fluoride toothpaste
- Placebo Oral Rinse (Placebo Comparator): Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 ml of Placebo Oral Rinse 2 for 1 minute. This regimen will be performed twice daily for 8 weeks.
  Interventions: Other: Placebo Oral Rinse; Drug: Standard fluoride toothpaste

INTERVENTIONS:
Device: Experimental Oral Rinse 1 — (1.5% w/w KOX, pH 4.5)
  Arms: Experimental Oral Rinse1
Device: Experimental Oral Rinse 2 — (1.5% w/w KOX, pH 7)
  Arms: Experimental Oral Rinse 2
Other: Placebo Oral Rinse — (0% w/w KOX, pH 4.5)
  Arms: Placebo Oral Rinse
Drug: Standard fluoride toothpaste — 1000ppm fluoride as sodium monofluorophosphate

SUMMARY:
This study will investigate the longitudinal efficacy of two experimental oral rinses containing 1.5% weight/weight (w/w) dipotassium oxalate monohydride (KOX), formulated at pH 4.5 and pH 7 respectively, for the relief of dentinal hypersensitivity (DH), compared to a placebo oral rinse, when used as an adjunct to twice daily brushing with a standard fluoride toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Aged between 18 and 55 years inclusive
* Good general and mental health with, in the opinion of the investigator or medically qualified designee:

A. No clinically significant and relevant abnormalities in medical history or upon oral examination.

B. Absence of any condition that would impact on the subject's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.

- Dental health

At Screening:

A. Self-reported history of dentinal hypersensitivity (DH) lasting more than six months but not more than 10 years.

B. Good general oral health, with a minimum of 20 natural teeth.

C. Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria:

* Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR).
* Tooth with modified gingival index (MGI) score =0 adjacent to the test area (exposed dentine) only and a clinical mobility of ≤1.
* Tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y/N response).

At Baseline:

D. Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), that meet all of the following criteria:

- Tooth with signs of sensitivity, measured by qualifying tactile stimulus (Yeaple ≤ 20g) and evaporative air assessment (Schiff Sensitivity Score ≥ 2)

Exclusion Criteria:

* Pregnant or breast feeding women
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain.
* Currently taking antibiotics or has taken antibiotics within two weeks of Baseline.
* Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia.
* Presence of kidney disease, hyperoxaluria, or any other condition that may be exacerbated by oxalic acid or oxalate salts.
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Any condition which, in the opinion of the investigator, causes xerostomia.
* Treatment of periodontal disease within 12 months of screening
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Recent history (within the last year) of alcohol or other substance abuse
* Dental prophylaxis within four weeks of Screening.
* Tongue or lip piercing or presence of dental implants.
* Desensitizing treatment within eight weeks of Screening (professional sensitivity treatments and non-toothpaste sensitivity treatments).
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening.
* Teeth bleaching within eight weeks of Screening
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening.
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.
* Sensitive tooth not expected to respond to treatment with an over-the-counter toothpaste in the opinion of the investigator.
* Use of an oral care product indicated for the relief of dentine hypersensitivity within eight weeks of screening
* Individuals who require antibiotic prophylaxis for dental procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 262 participants were screened, out of which 240 participants were randomized and 238 completed the study.
Groups:
- Experimental Oral Rinse 1: Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 mL of Experimental Oral Rinse 1 (1.5% weight by weight (w/w) dipotasium oxalate monohydrate [KOX], pH 4.5) for 1 minute. This regimen was performed twice daily for 8 weeks.
- Experimental Oral Rinse 2: Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 mL of Experimental Oral Rinse 2 (1.5% w/w KOX, pH 7) for 1 minute. This regimen was performed twice daily for 8 weeks.
- Placebo Oral Rinse: Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 mL of Placebo Oral Rinse (0% w/w KOX, pH 4.5) for 1 minute. This regimen was performed twice daily for 8 weeks.
Period: Overall Study
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Started | 79 | 80 | 81
Completed | 78 | 79 | 81
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Oral Rinse1: Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 mL of Experimental Oral Rinse 1 (1.5% w/w KOX, pH 4.5) for 1 minute. This regimen was performed twice daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Experimental Oral Rinse1 | Experimental Oral Rinse 2 | Placebo Oral Rinse | Total
Number analyzed (Participants) | 79 | 80 | 81 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (10.45) | 35.0 (8.41) | 36.5 (10.07) | 35.4 (9.67)
Gender [Count of Participants; unit: Participants]
  Female | 51 | 53 | 56 | 160
  Male | 28 | 27 | 25 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score of Experimental Oral Rinses 1 and 2 Against a Placebo Oral Rinse at Week 8
Description: The examiner assessed the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicate improvement in sensitivity.
Time Frame: Baseline, Week 8
Population: Intent-to-treat (ITT) population included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Oral Rinse1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 78 | 79 | 81
score on a scale
  At Baseline | 2.54 (0.420) | 2.56 (0.416) | 2.55 (0.415)
  Change from Baseline at Week 8 | -0.86 (0.772) | -0.66 (0.803) | -0.73 (0.779)
Statistical Analysis 1: Comparison: Experimental Oral Rinse1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.4350, ANCOVA — From ANCOVA model with treatment as factor and baseline Schiff score as covariate. For the Week 8 comparisons of the two test groups against the control group, Dunnett's multiplicity adjustment is applied; Least square (LS) mean difference = -0.13, 95% CI 2-sided [-0.400 to 0.134] — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment. For Week 8 comparisons of the two test groups against the control group, Dunnett's multiplicity adjustment is applied
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.7605, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.07, 95% CI 2-sided [-0.192 to 0.340] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score of Two Experimental Oral Rinses 1 and 2 at Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: ITT population included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Oral Rinse1 | Experimental Oral Rinse 2
Number analyzed (Participants) | 78 | 79
score on a scale
  At Baseline | 2.54 (0.420) | 2.56 (0.416)
  Change from Baseline at Week 8 | -0.86 (0.772) | -0.66 (0.803)
Statistical Analysis 1: Comparison: Experimental Oral Rinse1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.0873, ANCOVA — From ANCOVA model with treatment as factor and baseline Schiff score as covariate; LS mean difference = -0.21, 95% CI 2-sided [-0.445 to 0.031] — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment

3. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score of Two Experimental Oral Rinses 1 and 2 and a Placebo Oral Rinse at Week 4
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Oral Rinse 1: Brushing with fluoride toothpaste for 1 minute followed by rinsing with 10 mL of Experimental Oral Rinse 1 (1.5% w/w KOX, pH 4.5) for 1 minute. This regimen was performed twice daily for 8 weeks.
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 78 | 79 | 81
score on a scale
  At Baseline | 2.54 (0.420) | 2.56 (0.416) | 2.55 (0.415)
  Change from Baseline at Week 4 | -0.63 (0.701) | -0.56 (0.670) | -0.57 (0.732)
Statistical Analysis 1: Comparison: Experimental Oral Rinse 1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.4921, ANCOVA — From ANCOVA model with treatment as factor and baseline Schiff score as covariate; LS mean difference = -0.07, 95% CI 2-sided [-0.270 to 0.130] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.8728, ANCOVA — From ANCOVA model with treatment as factor and baseline Schiff score as covariate; LS mean difference = 0.02, 95% CI 2-sided [-0.183 to 0.216] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse 1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.4003, ANCOVA — From ANCOVA model with treatment as factor and baseline Schiff score as covariate; LS mean difference = -0.09, 95% CI 2-sided [-0.287 to 0.115] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Tactile Threshold (Gram [g]) of Two Experimental Oral Rinses 1 and 2 and a Placebo Oral Rinse at Week 4
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force has reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline, the maximum force used was 20g; at all subsequent visits, it was 80g. However, in situations where participants did not give a 'yes' response at force of 80g, the tactile threshold was recorded as >80g. For analysis purposes values recorded as >80g were treated as 90g values.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Median (Full Range); unit: g
Arm/Group | Experimental Oral Rinse1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 78 | 79 | 81
g
  At Baseline | 10.00 (0.000) [10.0 to 10.0] | 10.00 (0.000) [10.0 to 10.0] | 10.00 (0.000) [10.0 to 10.0]
  Change from Baseline at Week 4 | 5.00 (16.371) [0.0 to 80.0] | 0.00 (14.692) [0.0 to 70.0] | 5.00 (13.219) [0.0 to 55.0]
Statistical Analysis 1: Comparison: Experimental Oral Rinse1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.8106, Van Elteren test — From Van Elteren test; Median Difference (Net) = 0.00, 95% CI 2-sided [0.000 to 0.000] — Median difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment. From non-parametric Hodges-Lehmann estimations
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.1656, Van Elteren test — From Van Elteren test; Median Difference (Net) = 0.00, 95% CI 2-sided [-5.000 to 0.000] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.1419, Van Elteren test; Median Difference (Net) = 0.00, 95% CI 2-sided [0.000 to 5.000] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline in Tactile Threshold (g) of Two Experimental Oral Rinses 1 and 2 and a Placebo Oral Rinse at Week 8
Description: as for outcome 4
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Median (Full Range); unit: g
Arm/Group | Experimental Oral Rinse1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 78 | 79 | 81
g
  At Baseline | 10.00 [10.0 to 10.0] | 10.00 [10.0 to 10.0] | 10.00 [10.0 to 10.0]
  Change from Baseline at Week 8 | 7.50 [0.0 to 80.0] | 5.00 [0.0 to 80.0] | 5.00 [0.0 to 80.0]
Statistical Analysis 1: Comparison: Experimental Oral Rinse1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.5631, Van Elteren test — From Van Elteren test; Median Difference (Net) = 0.00, 95% CI 2-sided [0.000 to 5.000] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.8423, Van Elteren test — From Van Elteren test; Median Difference (Net) = 0.00, 95% CI 2-sided [0.000 to 0.000] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.4390, Van Elteren test — From Van Elteren test; Median Difference (Net) = 0.00, 95% CI 2-sided [0.000 to 5.000] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Change From Baseline in Visual Rating Scale (VRS) of Two Experimental Oral Rinses 1 and 2 and a Placebo Oral Rinse) at Week 4
Description: Participants rated the intensity of their response to the evaporative (air) stimulus using a 10 point VRS. The Participants were asked to rate their pain on a scale of 1 ("No Pain") to 10 ("Intense Pain"). A reduction in the score is indicative of an improvement in sensitivity.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Oral Rinse1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 78 | 79 | 81
score on a scale
  At Baseline | 6.22 (1.515) | 6.32 (1.209) | 6.19 (1.422)
  Change from Baseline at Week 4 | -1.60 (1.476) | -1.29 (1.669) | -1.45 (1.505)
Statistical Analysis 1: Comparison: Experimental Oral Rinse1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.5170, ANCOVA — From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline VRS as covariate; LS mean difference = -0.15, 95% CI 2-sided [-0.611 to 0.308] — From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline VRS as covariate. Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.4538, ANCOVA — From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline VRS as covariate; LS mean difference = 0.17, 95% CI 2-sided [-0.284 to 0.633] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.1663, ANCOVA — From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline VRS as covariate; LS mean difference = -0.33, 95% CI 2-sided [-0.788 to 0.136] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline in VRS of Two Experimental Oral Rinses 1 and 2 and a Placebo Oral Rinse) at Week 8
Description: as for outcome 6
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Oral Rinse1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Number analyzed (Participants) | 78 | 79 | 81
score on a scale
  At Baseline | 6.22 (1.515) | 6.32 (1.209) | 6.19 (1.422)
  Change from Baseline at Week 8 | -2.25 (1.781) | -2.07 (1.820) | -2.15 (1.865)
Statistical Analysis 1: Comparison: Experimental Oral Rinse1 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.7137, ANCOVA — From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline VRS as covariate; LS mean difference = -0.10, 95% CI 2-sided [-0.661 to 0.453] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Experimental Oral Rinse 2 vs Placebo Oral Rinse; Test type: Superiority or Other; p = 0.7353, ANCOVA — From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline VRS as covariate; LS mean difference = 0.10, 95% CI 2-sided [-0.460 to 0.651] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Experimental Oral Rinse1 vs Experimental Oral Rinse 2; Test type: Superiority or Other; p = 0.4843, ANCOVA — From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline VRS as covariate; LS mean difference = -0.20, 95% CI 2-sided [-0.760 to 0.361] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Arm/Group | Experimental Oral Rinse 1 | Experimental Oral Rinse 2 | Placebo Oral Rinse
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/80 | 0/81
Other Adverse Events (participants affected / at risk) | 11/79 | 13/80 | 11/81
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Oral Rinse 1 (N=79) | Experimental Oral Rinse 2 (N=80) | Placebo Oral Rinse (N=81)
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 5 | 7 | 8
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 3 | 2 | 0
DENTAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 1 | 0 | 1
CHAPPED LIPS (Gastrointestinal disorders) | 0 | 0 | 1
LEUKOPLAKIA ORAL (Gastrointestinal disorders) | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 2 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1 | 1
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.